CLINICAL TRIAL: NCT00816920
Title: Diagnosis and Evolution of Isolated Deep Vein Thrombosis of the Calf in Symptomatic Outpatients. The Blind, Prospective "CALTHRO" Study.
Brief Title: Natural History of Isolated Deep Vein Thrombosis of the Calf
Acronym: CALTHRO
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: 24/2001/O EM60/2007/O
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Isolated Distal DVT; Proximal DVT; Pulmonary Embolism
Keywords: distal DVT; calf DVT; DVT diagnosis; management of patients with suspected leg DVT
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Outpatients with suspected leg DVT after exclusion of proximal DVT
  Interventions: Other: Ultrasound examination of leg veins

INTERVENTIONS:
Other: Ultrasound examination of leg veins — Outpatients symptomatic for leg DVT follow the standard diagnostic procedure (ultrasound examination of proximal deep veins, pre-test clinical probability and D-dimer, and a second US after 5-7 days) to exclude proximal DVT; they also receive by another doctor a complete US examination of the deep leg veins to assess the presence of isolated calf DVT, the results of the latter examination are kept blind to the patient and to the treating doctor, and disclosed after three months

SUMMARY:
Whether isolated distal DVT (IDDVT), DVT confined to the calf, should be looked for and diagnosed to allow them to be treated with anticoagulants remains one of the still unsolved issues in vascular medicine, especially because of the insufficient data on clinical risks of untreated distal DVT. Management studies have shown that it is safe to withhold anticoagulation in outpatients with suspected DVT if compression ultrasonography (CUS) limited to the proximal deep veins yields normal results on presentation and on repeated examination after 5 to 7 days. This strategy is based on the premise that IDDVT do not need to be diagnosed and treated, what is necessary when they extend involving the proximal veins. There is no general agreement, however, on the assumption that the non-extending IDDVT do not need to be diagnosed and treated, and many authors recommend to perform a single CUS examination extended to the distal deep veins. All the available studies have treated with anticoagulants the diagnosed IDDVT and no adequate information is available on the risk of IDDVT left untreated.

The present study, performed in outpatients with suspected leg DVT, aims at assessing the clinical consequences of IDDVT diagnosed (by a complete US investigation) but not treated because the results of this investigation remain blind to both the patient and the treating doctor, whereas the diagnostic-therapeutic procedure remains the usual one, based on CUS investigation limited to diagnose proximal DVT, to be repeated after 5-7 days (or earlier) to exclude an extension to proximal veins of an IDDVT potentially present.

DETAILED DESCRIPTION:
Outpatients symptomatic for suspected DVT of a leg are examined by a vascular doctor according to standard procedure based on pre-test clinical probability (PTCP) assessment, D-dimer assay and a CUS limited to the proximal deep veins. Those in whom a proximal DVT is excluded and have intermediate/high PTCP or altered D-dimer level are eligible for the study. The included patients are immediately submitted to an extensive echo-color-Doppler examination of calf deep veins by a different vascular doctor and results are closed in an envelope that will be open after three months (or before if necessary). In the meantime, patients will follow the standard diagnostic procedure: they receive an appointment to come back in 5-7 days for a further CUS examination, or even before in case of worsening of symptoms/signs. All the included patients receive a telephone call after three months to exclude possible complications.

ELIGIBILITY:
Inclusion Criteria:

* suspected deep vein thrombosis of a leg
* intermediate/high pre-test clinical probability or high D-dimer levels

Exclusion Criteria:

* age < 18 years
* presence of proximal DVT
* suspected isolated iliac DVT
* symptoms/signs lasting from > 30 days
* presence of symptoms of pulmonary embolism
* pregnancy or puerperium
* full dose treatment with heparin or derivatives from > 1 day
* presence of superficial vein thrombosis
* limited life expectancy (< 6 months)
* geographically inaccessible location
* inability or refusal to give consent
* participation in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients with suspected deep vein thrombosis (DVT) of a leg in whom a proximal DVT is excluded.
  The study is not funded. As a result, it will not be possible to enroll all consecutive eligible patients; rather patients will be included based on the availability of expert medical staff in the day of their presentation (in general the first patient of the day).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Thrombotic complications (deep vein thrombosis and/or pulmonary embolism within three months from first examination | three months from first examination

SECONDARY OUTCOMES:
other vascular complications; how many isolated distal DVT will be diagnosed | three months from first examination

CONTACTS AND LOCATIONS:
Overall Officials: Gualtiero Palareti, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Bologna, Policlinico S. Orsola-Malpighi
Locations (2):
- Italy (2):
  - Angiology & Blood Coagulation, Policlinico S. Orsola-Malpighi, Bologna
  - Servizio di Fisiopatologia Vascoalre, Casa di Cura Villa Serena, Pescara